CLINICAL TRIAL: NCT02745509
Title: A Prospective, Multicentral, Open-label, Randomized, Controlled Clinical Trial to Investigation the Value of Extensive Intraoperative Peritoneal Lavage After Curative Gastrectomy for Locally Advanced Gastric Cancer
Brief Title: Extensive Intraoperative Peritoneal Lavage After Curative Gastrectomy for Locally Advanced Gastric Cancer (SEIPLUS)
Acronym: SEIPLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Anqing Municipal Hospital (Other); Yuebei People's Hospital (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Jiangsu Cancer Institute & Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Affiliated Hospital of Wannan Medical College (Other); Lishui hospital of Zhejiang University (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Study Chair, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEIPLUS
Record Dates: First submitted 2016-03-28; First posted 2016-04-20 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Gastric Cancer
Keywords: Extensive Intraoperative Peritoneal Lavage; EIPL; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extensive Intraoperative Peritoneal Lavage (Experimental): Gastrectomy with D2 lymphadenectomy is performed. The peritoneal cavity of subject will be washed with 10 liters of warmed normal saline (1 liter per cycle for 10 cycles), followed by complete aspiration of the fluid . The abdomen will be closed as per standard.
  Interventions: Other: Extensive Intraoperative Peritoneal Lavage
- Standard Treatment (No Intervention): Gastrectomy with D2 lymphadenectomy is performed. The peritoneal lavage will be done < 3 cycles with 3 liters or less of warmed normal saline. The abdomen will be closed as per standard.

INTERVENTIONS:
Other: Extensive Intraoperative Peritoneal Lavage — Extensive Intraoperative Peritoneal Lavage
  Other Names: EIPL
  Arms: Extensive Intraoperative Peritoneal Lavage

SUMMARY:
The investigators study aims to explore the potential function of extensive intraoperative peritoneal lavage in improving the overall survival and progression-free survival for locally advanced gastric cancer after curative resection.

Hypothesis: Overall survival and progression-free survival of locally advanced gastric cancer are improved by extensive intraoperative peritoneal lavage.

DETAILED DESCRIPTION:
Gastric cancer has been one of the most frequently common cancers and remains the third leading cause of death among malignant tumors all over the world. Surgery has always been considered as the most effective treatment. While significant surgical technique and perioperative management have dramatically improved the survival of patients with advanced gastric cancer, patients with T4 stage or serosal-positive gastric cancer often suffer from recurrence as peritoneal dissemination, and the prognosis of those patients is extremely poor. Despite curatively resected, Peritoneal metastasis is completed by the implantation of peritoneal free cancer cells exfoliated from serosa-invasive tumors. Therefore, things need to be done to eliminate the free exfoliated cancer cells on the peritoneal lining in order to reduce the risk of peritoneal recurrence.

A multi-institutional prospective, randomized trial has been launched by Kuramoto recently. The trail was intended to demonstrate the superiority in overall survival of addition of Extensive Intraoperative peritoneal Lavage (EIPL) to standard treatment in patients with≥T3 carcinoma of stomach. Based on the'limiting dilution theory', after total or distal gastrectomy with D2 lymphadenectomy, the peritoneal cavity is extensively rinsed 10 times with 1 L physiological saline at a time, followed by complete aspiration of the fluid. In total, 10 L saline is to be used. In this study, the EIPL-IPC group had a significantly lower incidence of peritoneal recurrence. Furthermore, the 5-year overall survival rate of the patients in the EIPL-IPC group (43.8%) was significantly better than that of the intraperitoneal chemotherapy (IPC) group (4.6%) and the surgery-alone group (0%). All in all, EIPL is easy to carry out, safe and inexpensive. Therefore, gastrectomy with EIPL will be a new standard treatment of gastric cancer.

To ensure the quality of the study, two interim analyses will be planned at the half and the completion of the study respectively. The Data and Safety Monitoring Committee will independently review the interim analysis and stop the study ahead of schedule if necessary. Furthermore, to improve the study progress and quality, the in-house interim monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old.
2. ECOG score standard (ECOG）performance status of 0 or 1 and expected to survive more than 6 months.
3. Without any other malignancies.
4. Written informed consent from the patient.
5. Histologically proven primary gastric adenocarcinoma.
6. Patients planned for open gastrectomy.
7. Patients who have T3 (subserosal) or T4 (serosal) disease based on Ultrasound gastroscopy and intra-operative inspection with any N staging and M0 gastric cancer.
8. No preoperative neoadjuvant chemotherapy.
9. Length of esophageal invasion≤3cm and no need of thoracotomy for resection.
10. Intraoperative inclusion criteria:

    1. Clinically T3, T4a or T4b.
    2. Clinically H0 and M0. No peritoneal dissemination or Distant metastases.
    3. Possible for R0 surgery.

Exclusion Criteria:

1. Female in pregnancy or lactation.
2. Supraclavicular lymph nodes metastases，pelvis or ovarian implantation，peritoneal dissemination，liver，lung and bone metastases.
3. Massive ascites or cachexia.
4. Patients participating in any other clinical trails currently，or participated in other trails within 1 months.
5. Without a history of stomach or esophageal cancers, including stromal tumor，sarcoma，lymphoma and carcinoid.
6. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases.
7. Patients with poor compliance or considered to be poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2016-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3-year
  The survival rate between the surgery to the 3rd year due to all-cause death or last follow-up.

SECONDARY OUTCOMES:
Disease-free survival | 3-year
  The progression-free or all-cause death rate between the surgery and the 3rd year.
Peritoneal recurrence | 3-year
  The Peritoneal recurrence rate between the surgery and the 3rd year
Postoperative complications | an average of 10 days
  complications such bleeding, infection, obstruction and leakage
Post-operative quality of life | an average of 10 days
  The postoperative quality of life will be assessed by factors such as Swallowing，Pain and discomfort，Dietary restrictions, Upper gastrointestinal symptoms, mental status and others.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Guangzhou, Guangdong
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Lishui Hospital of Zhejiang University, Lishui, Zhejiang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mezhir JJ, Posner MC, Roggin KK. Prospective clinical trial of diagnostic peritoneal lavage to detect positive peritoneal cytology in patients with gastric cancer. J Surg Oncol. 2013 Jun;107(8):794-8. doi: 10.1002/jso.23328. Epub 2013 Mar 26. PMID 23532564
- [Background] Tang B, Peng ZH, Yu PW, Yu G, Qian F, Zeng DZ, Zhao YL, Shi Y, Hao YX, Luo HX. Aberrant expression of Cx43 is associated with the peritoneal metastasis of gastric cancer and Cx43-mediated gap junction enhances gastric cancer cell diapedesis from peritoneal mesothelium. PLoS One. 2013 Sep 11;8(9):e74527. doi: 10.1371/journal.pone.0074527. eCollection 2013. PMID 24040271
- [Background] Hamazoe R, Maeta M, Kaibara N. Intraperitoneal thermochemotherapy for prevention of peritoneal recurrence of gastric cancer. Final results of a randomized controlled study. Cancer. 1994 Apr 15;73(8):2048-52. doi: 10.1002/1097-0142(19940415)73:83.0.co;2-q. PMID 8156509
- [Background] Xu DZ, Zhan YQ, Sun XW, Cao SM, Geng QR. Meta-analysis of intraperitoneal chemotherapy for gastric cancer. World J Gastroenterol. 2004 Sep 15;10(18):2727-30. doi: 10.3748/wjg.v10.i18.2727. PMID 15309728
- [Background] Sautner T, Hofbauer F, Depisch D, Schiessel R, Jakesz R. Adjuvant intraperitoneal cisplatin chemotherapy does not improve long-term survival after surgery for advanced gastric cancer. J Clin Oncol. 1994 May;12(5):970-4. doi: 10.1200/JCO.1994.12.5.970. PMID 8164049
- [Background] Rosen HR, Jatzko G, Repse S, Potrc S, Neudorfer H, Sandbichler P, Zacherl J, Rabl H, Holzberger P, Lisborg P, Czeijka M. Adjuvant intraperitoneal chemotherapy with carbon-adsorbed mitomycin in patients with gastric cancer: results of a randomized multicenter trial of the Austrian Working Group for Surgical Oncology. J Clin Oncol. 1998 Aug;16(8):2733-8. doi: 10.1200/JCO.1998.16.8.2733. PMID 9704725
- [Background] Coccolini F, Cotte E, Glehen O, Lotti M, Poiasina E, Catena F, Yonemura Y, Ansaloni L. Intraperitoneal chemotherapy in advanced gastric cancer. Meta-analysis of randomized trials. Eur J Surg Oncol. 2014 Jan;40(1):12-26. doi: 10.1016/j.ejso.2013.10.019. Epub 2013 Nov 5. PMID 24290371
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Yagi Y, Matsuda M, Yonemura Y, Baba H. Extensive intraoperative peritoneal lavage as a standard prophylactic strategy for peritoneal recurrence in patients with gastric carcinoma. Ann Surg. 2009 Aug;250(2):242-6. doi: 10.1097/SLA.0b013e3181b0c80e. PMID 19638909
- [Background] Misawa K, Mochizuki Y, Ohashi N, Matsui T, Nakayama H, Tsuboi K, Sakai M, Ito S, Morita S, Kodera Y. A randomized phase III trial exploring the prognostic value of extensive intraoperative peritoneal lavage in addition to standard treatment for resectable advanced gastric cancer: CCOG 1102 study. Jpn J Clin Oncol. 2014 Jan;44(1):101-3. doi: 10.1093/jjco/hyt157. Epub 2013 Nov 27. PMID 24287077
- [Derived] Guo J, Xu A, Sun X, Zhao X, Xia Y, Rao H, Zhang Y, Zhang R, Chen L, Zhang T, Li G, Xu H, Xu D. Three-year outcomes of the randomized phase III SEIPLUS trial of extensive intraoperative peritoneal lavage for locally advanced gastric cancer. Nat Commun. 2021 Nov 15;12(1):6598. doi: 10.1038/s41467-021-26778-8. PMID 34782599
- [Derived] Guo J, Xu A, Sun X, Zhao X, Xia Y, Rao H, Zhang Y, Zhang R, Chen L, Zhang T, Li G, Xu H, Xu D. Combined Surgery and Extensive Intraoperative Peritoneal Lavage vs Surgery Alone for Treatment of Locally Advanced Gastric Cancer: The SEIPLUS Randomized Clinical Trial. JAMA Surg. 2019 Jul 1;154(7):610-616. doi: 10.1001/jamasurg.2019.0153. PMID 30916742
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html
- See also: Stomach Cancer — http://www.nlm.nih.gov/medlineplus/stomachcancer.html
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks